CLINICAL TRIAL: NCT00947102
Title: Observational Study - Influence of Gemcitabine Treatment on Immunological and Serological Profile in Patients With Pancreatic Tubular Carcinoma
Brief Title: Influence of Gemcitabine Treatment on Immunological and Serological Profile in Patients With Pancreatic Cancer
Acronym: GEMSTHER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Blood Transfusion Centre of Slovenia (Other Government)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Primoz Rozman MD, PhD, Blood Transfusion Centre of Ljubljana
Other Study IDs: Gemcitabine1
Record Dates: First submitted 2009-07-24; First posted 2009-07-27 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-07

CONDITIONS: Pancreatic Tubular Adenocarcinoma
Keywords: pancreatic tubular adenocarcinoma; gemcitabine; gene expression; immunological status; serological status; pancreatic tubular adenocarcinoma adjuvant setting
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic tubular adenocarcinoma: Patients with pancreatic tubular adenocarcinoma
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation

SUMMARY:
Observational study of influence of gemcitabine treatment on serological and immunological status and gene expression profile in patients with pancreatic tubular carcinoma after tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-2 at the time of inclusion
* Following R0 or R1 pancreatic tubular adenocarcinoma resection

Exclusion Criteria:

* Pregnancy
* Serious comorbidity

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after resection of pancreatic tubular adenocarcinoma
Sampling Method: Non-Probability Sample
Dates: Start 2009-02; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana; Department for Gastroenterology, Ljubljana, Ljubljana, Slovenia